CLINICAL TRIAL: NCT06050187
Title: Accuracy of 3-dimensional Printed Implant Cast Versus Conventional Stone Cast for Edentulous Mandibular Arch: A Comparative Study
Brief Title: Accuracy of 3-dimensional Printed Implant Cast Versus Conventional Stone Cast for Edentulous Mandibular Arch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A07030123
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-09

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I conventional stone cast (Active Comparator): Mandibular stone cast with 4 parallel implants analogues in canines and second premolar regions will be fabricated conventionally.
  Interventions: Procedure: implant casts fabrication
- Group II 3D printed implant cast (Active Comparator): 3D printed implant mandibular cast with 4 parallel digital implants analogues in canines and second premolar regions will be fabricated digitally.
  Interventions: Procedure: implant casts fabrication

INTERVENTIONS:
Procedure: implant casts fabrication — four implant casts fabricated

SUMMARY:
This study will be conducted to compare between accuracy of 3D printed implant cast produced from digital impression and conventional stone cast produced from conventional splinted open tray impression for edentulous mandibular arch with four implants.

ELIGIBILITY:
Inclusion Criteria:

* • Patients were healthy and free from all systemic diseases that affect osseointegration or bone resorption around the implant as recorded from medical and dental history.

  * Patients were free from all oral pathological conditions and any remaining roots which were verified by pre-operative panoramic radiograph.
  * Patients with U shaped arch, flat mandibular alveolar ridge covered with even compressibility healthy mucosa and gingival thickness of about 2mm verified by dual scan of cone beam computed tomography (CBCT) during treatment planning. Fig.(1)
  * Adequate residual alveolar bone quality D2 bone type in the anterior and premolar regions according to the Misch bone density classification scheme (850 to1250 housefield units) confirmed by CBCT.
  * Angel's class I maxillomandibular relation with moderate inter- arch space (20 mm) confirmed through tentative jaw relationship, and restorative space of at least 15 mm determined by putty index technique
  * Patients complain from poor retentive mandibular denture seeking for alternative fixed options.
  * Patient who is motivated, agreed with the follow-up visits and willing to return for follow-up appointments.

Exclusion Criteria:

* • Patient with absolute contraindications that interfere with surgical placement and osseointegration of implants as uncontrolled diabetes mellitus, generalized osteoporosis, recent myocardial infarction, patient with radiotherapy.

  * Patient with relative contraindication such as UN controlled diabetes mellitus, moderate smoking and alcoholism, patient with TMJ disorder and heavy smokers for more than10 cigarettes per day.
  * Patient with local contra indication as insufficient bone quality, localized lesion in canine area and premolar area, unfavourable position of the lower alveolar or mental nerve, bone defects as verified by cone beam CT.
  * Uncooperative patient.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-12-27 (Estimated); Study Completion 2024-12-17 (Estimated)

PRIMARY OUTCOMES:
accuracy of 3D printed casts | 6 month
  Accuracy of 3D printed casts will be evaluated digitally by geomagic software

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No